CLINICAL TRIAL: NCT06665997
Title: Clinical and Biomarker Effects of Depot Medroxyprogesterone Acetate in Females With Sickle Cell Disease
Acronym: SCD Depo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Emory University (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Andrea Roe, MD, MPH, Assistant Professor of Obstetrics and Gynecology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 857039; 1R01HL175726-01 (NIH)
Record Dates: First submitted 2024-10-23; First posted 2024-10-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease (SCD); Vaso-Occlusive Pain Episode in Sickle Cell Disease
Keywords: Sickle Cell Disease; Depot Medroxyprogesterone Acetate (Depo-Provera); Contraception; Vaso-Occlusive Pain
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Depot Medroxyprogesterone Acetate (Depo-Provera) (Experimental): All participants will receive a 150mg dose intramuscular administration of depot medroxyprogesterone acetate (DMPA) injectable suspension after a 3-month baseline with no hormonal contraception.
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate (DMPA) — 150mg dose intramuscular administration of depot medroxyprogesterone acetate (DMPA) injectable suspension

SUMMARY:
This research is being conducted to see if using an injectable contraception, Depot Medroxyprogesterone Acetate (Depo-Provera), can reduce the pain experienced by women with sickle cell disease.

Participants in this study will be adult women with sickle cell disease who regularly experience sickle cell pain. They will complete a 3-month "baseline "with no use of hormonal contraception, and then a 3-month follow-up after receiving an injection of Depo-Provera. Participants will complete 6 to 7 in-person visits with a urine pregnancy test, blood draw, and surveys, as well as complete remote weekly surveys and monthly home pregnancy tests.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Female, aged 18-50 years old
3. Diagnosis of sickle cell disease (SS, SB0,SB+,SC)
4. Report of at least 1 vaso-occlusive pain episode per month on average in the previous 6 months
5. At least 1 and no more than 10 medical presentations (e.g. hospitalization, emergency room visit, outpatient infusion visit) for sickle cell-related pain during the past year
6. Willing to discontinue any hormonal contraception at the time of enrollment. Washout period of 1 month since last use of all hormonal contraception, and 4 months since most recent administration of depot medroxyprogesterone, is required prior to enrollment in the study.
7. Have regular menstrual cycles (when not on hormonal contraception) with a usual length of 21 to 35 days.
8. Stable dose of hydroxyurea and other sickle cell-related medications for the past 6 months
9. Access to a device with text-messaging capability
10. Must be able to read and understand English
11. Willing to comply with study procedures

Exclusion Criteria:

1. Chronic inflammatory conditions, such as lupus or inflammatory bowel disease
2. History of VTE or stroke
3. Current use of crizanlizumab, voxelotor, or red cell exchange transfusion, or history of hematopoietic stem cell transplantation
4. Current use of hormonal contraception or the copper intrauterine device
5. Current pregnancy or pregnancy within the last 6 months
6. Current lactation
7. Polycystic ovary syndrome or irregular periods
8. Blood pressure >= 160 systolic or >=100 diastolic at screening visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute vaso-occlusive episodes | 6 months
  The primary outcome is frequency of VOEs during each phase (baseline and intervention). A VOE is self-reported by the participant. Discrete pain episodes will be separated by at least 2 weeks from one other.
  During both the baseline and intervention study phases, participants will provide weekly reports via electronic survey of vaso-occlusive pain. VOE will be defined as self-reported typical SCD pain that interferes with usual daily activities or requires emergency care or hospitalization, with distinct episodes separated by at least 2 weeks without pain.

SECONDARY OUTCOMES:
C-reactive protein | 6 months
  C-reactive protein will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
Hemoglobin | 6 months
  Hemoglobin will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
Reticulocyte count | 6 months
  Reticulocyte count will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
Platelet count | 6 months
  Platelet count will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
Fetal hemoglobin | 6 months
  Fetal hemoglobin will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
Bilirubin | 6 months
  Bilirubin will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
D-dimer | 6 months
  D-dimer will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).
von Willebrand factor | 6 months
  von Willebrand factor will be measured from blood samples drawn twice, once during each study phase (baseline and intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Roe, MD MPH, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) for use by other researchers including those outside of the study.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be made available starting 6 months after publication. There is no planned end date.
Access Criteria: Researchers will obtain access through NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) in accordance with their SOPs.
URL: https://biolincc.nhlbi.nih.gov/